CLINICAL TRIAL: NCT02103270
Title: Single Center, Placebo Controlled Clinical Study in Desensitization vs Tolerance Induction in Peanut Allergy Subjects
Brief Title: The Peanut Oral Immunotherapy Study: Safety, Efficacy and Discovery
Acronym: POISED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kari Christine Nadeau, MD PhD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: AADCRC-STAN-001
Record Dates: First submitted 2014-03-25; First posted 2014-04-03 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oat Flour 600 mg (Placebo Comparator): Arm C that is maintained on placebo (oat flour) throughout the study; this arm will receive 600 mg oat flour beginning on week 104. This will be true even if a subject in the placebo group meets criteria at week 104
  Interventions: Drug: Oat Flour
- Peanut Protein 4,000mg (Active Comparator): Arm A on peanut OIT until week 104 (maintenance) and once meeting criteria [i.e. 1) on OIT treatment for minimum 104 weeks, 2) taking daily maintenance dose of 4,000 mg protein for at least 13 weeks, 3) no severe reactions to home dosing from Week 91-Week 104, and 4) no reactions at the Week 104 DBPCFC] will be assigned to avoid peanut (i.e. will consume 600 mg oat flour daily) and will proceed to tolerance and desensitization phase.
  Interventions: Drug: Peanut Protein 4,000mg; Drug: Oat Flour
- Peanut Protein 300 mg (Active Comparator): Arm B on peanut OIT until week 104 and once meeting criteria specified in description of Arm A, will be assigned to be maintained on 300 mg peanut protein (i.e. 600 mg peanut flour) daily and will proceed to the tolerance and desensitization testing phase.
  Interventions: Drug: Oat Flour; Drug: Peanut Protein 300 mg

INTERVENTIONS:
Drug: Peanut Protein 4,000mg — Arm A will be defined as "clinically tolerant" if there is no clinical reactivity at the Week 104 and Week 117 DBPCFC. Clinical reactivity is defined as any reaction ≥ Grade 1 based on the Bock's Criteria (Appendix 4). Individuals in Arm A who meet the definition of "clinically tolerant" will continue to avoid peanut protein (i.e. continue on 600 mg per day of oat flour) as long as each subsequent DBPCFC (performed every 13 weeks until end of study) shows no clinical reactivity.
  Other Names: Peanut Flour
  Arms: Peanut Protein 4,000mg
Drug: Oat Flour — Arm C will be defined as "natural loss of responsiveness" if they show no clinical reactivity at DBPCFCs (week 117 to end of study).
Drug: Peanut Protein 300 mg — Arm B will be defined as "desensitized" to a minimum of 300 mg per day of peanut protein if they show no clinical reactivity at DBPCFCs (week 117 to end of study).
  Other Names: Peanut Flour
  Arms: Peanut Protein 300 mg

SUMMARY:
Determine whether peanut oral immunotherapy (OIT) induces clinical tolerance as assessed after the initial 3 month avoidance period

Secondary Objectives:

* Identify the basic immune mechanisms which can explain the differences in the effects of OIT in desensitized vs. tolerant individuals.
* Determine whether immune monitoring measurements reflecting underlying mechanisms during OIT can be used to predict responses to OIT in individual subjects and, ultimately, to improve the safety and efficacy outcomes in peanut OIT protocols.

DETAILED DESCRIPTION:
All arms will undergo an Initial Dose Escalation (IDE) Day and updosing regimen with a maintenance phase of OIT or placebo to a maximum of 4,000 mg protein daily, as peanut flour, in the OIT groups, and to a maximum of an equivalent amount of oat flour for the placebo group. After maintenance is achieved, all subjects will begin performing DBPCFCs (staged so as to ensure safety) at Week 104 and every 13 weeks thereafter. At Week 104, individuals that reach criteria will, based on the randomization that was done at the start of the study, either stop therapy with peanut and be switched to oat flour, or will be maintained on 300 mg peanut protein per day and all placebo subjects will decrease to the equivalent volume of oat flour (approximately 600 mg oat flour) to optimize the blind. All subjects will be evaluated every 13 weeks thereafter with DBPCFCs until the end of study.

Individuals in Arm A will be defined as "clinically tolerant" if there is no clinical reactivity at the Week 104 and Week 117 DBPCFC. Clinical reactivity is defined as any reaction ≥ Grade 1 based on the Bock's Criteria. Individuals in Arm A who meet the definition of "clinically tolerant" will continue to avoid peanut protein (i.e. continue on 600 mg per day of oat flour) as long as each subsequent DBPCFC (performed every 13 weeks until end of study) shows no clinical reactivity.

Individuals in Arm B will be defined as "desensitized" to a minimum of 300 mg per day of peanut protein if they show no clinical reactivity at DBPCFCs (week 117 to end of study).

Individuals in Arm C will be defined as "natural loss of responsiveness" if they show no clinical reactivity at DBPCFCs (week 117 to end of study).

We plan to identify the basic immune mechanisms which can explain the differences in the effects of OIT in individuals who do or do not become clinically tolerant and to determine whether immune monitoring can predict the safety and efficacy outcomes in peanut OIT protocols.

After initial screening and enrollment, there are three phases of the study:

* Dose escalation and Build up Phase
* Maintenance phase
* Tolerance and Desensitization Testing phase Overall, 120 subjects who are eligible will undergo the Initial Dose Escalation Day. Subsequent updosing visits will occur every 2 weeks as a part of the build-up phase. They will continue to updose until they reach 4,000 mg protein daily, which is the maximum maintenance amount of protein. We expect active OIT treatment subjects to reach 4,000 mg of peanut protein between 44-78 weeks.

Treatment and Desensitization Failures:

A treatment failure will be defined as a) failure to reach 1.5 mg peanut protein (single dose) during the Initial Dose Escalation Day or b) failure to reach 1,000 mg peanut protein by week 104.

Subjects who do not meet the criteria at Week 104 and who demonstrate clinical reactivity will be considered desensitization failures.

If Arm B subjects demonstrate clinical reactivity in any DBPCFC from Week 117 to end of study, they will be considered desensitization failures.

If Arm A subjects demonstrate clinical reactivity (≥Grade 1, in any DBPCFC from Week 117 to end of study, they will be considered tolerance failures.

Treatment failures, desensitization failures, and tolerance failures will be unblinded (both participant and research staff) and will be followed until the end of the study at the specified study visits but will not undergo DBPCFCs. They will be considered in statistical analyses of the intent-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian must be able to understand and provide informed consent and/or assent as applicable.
* Peanut-allergic subjects between the ages of 7-55 years old.
* Sensitivity to peanut allergen as documented by a positive skin prick test result (5 mm or greater diameter wheal relative to negative control) within 10 months preceding enrollment.
* Allergy to peanut based on a double-blind placebo-controlled oral food challenge (DBPCFC) (see Appendix 4 for scoring details) failed at a dose ≤500 mg with peanut protein within 10 months preceding enrollment.
* All female subjects of child-bearing potential will be required to provide a blood or urine sample for pregnancy testing that must be negative one week before being allowed to participate in the study.
* Subjects must plan to remain in the study area during the trial.
* Subjects must be trained on the proper use of the EpiPen (see Appendix 6) to be allowed to enroll in the study.
* Subjects with other food allergies must agree to eliminate these other food items from their diet so as not to confound the safety and efficacy data from the study.
* Use of birth control by female subjects of child-bearing potential

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* History of cardiovascular disease
* History of other chronic disease (other than asthma, atopic dermatitis, or rhinitis) requiring therapy (e.g., heart disease, diabetes) that, in the opinion of the Principal Investigator, would represent a risk to the subject's health or safety in this study or the subject's ability to comply with the study protocol
* History of eosinophilic gastrointestinal disease
* Current participation in any other interventional study
* Subject is on 'build-up phase" of immunotherapy to another allergen (i.e., has not reached maintenance dosing)
* Severe asthma (2007 NHLBI Criteria Steps 5 or 6) at time of enrollment
* • Use of complementary and alternative medicine (CAM) treatment modalities (e.g., herbal remedies) for atopic and/or non-atopic disease within 90 days preceding Initial Dose Escalation Day (IDED) or at any time after the IDED
* Inability to discontinue antihistamines for the initial day of escalation, skin testing or OFCs
* Use of omalizumab within the past six months, or current use of other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator therapy (not including corticosteroids)
* Use of β-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Pregnancy or lactation
* History of sensitivity to oat
* History of severe anaphylaxis to peanut with symptoms including hypotension requiring fluid resuscitation and/or the need for mechanical ventilation
* Use of investigational drugs within 24 weeks of participation
* Past or current medical problems or findings from physical assessment or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari C Nadeau, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Sean N. Parker Center for Allergy Research at Stanford University, Mountain View, California, United States

REFERENCES:
- [Derived] Kanchan K, Cerosaletti K, Perry JA, DuToit G, Manohar M, Ling H, Paschall JE, Sanda S, Chinthrajah RS, Nepom GT, Nadeau KC, Jones SM, Lack G, Ruczinski I, Mathias RA. Genetic Determinants of Peanut-Specific IgG4 Levels in the Context of Sustained Oral Peanut Exposure in the LEAP Study. Immunology. 2026 Jan 30. doi: 10.1111/imm.70098. Online ahead of print. PMID 41615410
- [Derived] Wang W, Lyu SC, Ji X, Gupta S, Manohar M, Dhondalay GKR, Chinthrajah S, Andorf S, Boyd SD, Tibshirani R, Galli SJ, Nadeau KC, Maecker HT. Transcriptional changes in peanut-specific CD4+ T cells over the course of oral immunotherapy. Clin Immunol. 2020 Oct;219:108568. doi: 10.1016/j.clim.2020.108568. Epub 2020 Aug 9. PMID 32783912
- [Derived] Wright BL, Fernandez-Becker NQ, Kambham N, Purington N, Cao S, Tupa D, Zhang W, Sindher SB, Rank MA, Kita H, Katzka DA, Shim KP, Bunning BJ, Doyle AD, Jacobsen EA, Tsai M, Boyd SD, Manohar M, Chinthrajah RS. Gastrointestinal Eosinophil Responses in a Longitudinal, Randomized Trial of Peanut Oral Immunotherapy. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1151-1159.e14. doi: 10.1016/j.cgh.2020.05.019. Epub 2020 May 17. PMID 32434067
- [Derived] Chinthrajah RS, Purington N, Andorf S, Long A, O'Laughlin KL, Lyu SC, Manohar M, Boyd SD, Tibshirani R, Maecker H, Plaut M, Mukai K, Tsai M, Desai M, Galli SJ, Nadeau KC. Sustained outcomes in oral immunotherapy for peanut allergy (POISED study): a large, randomised, double-blind, placebo-controlled, phase 2 study. Lancet. 2019 Oct 19;394(10207):1437-1449. doi: 10.1016/S0140-6736(19)31793-3. Epub 2019 Sep 12. PMID 31522849
- [Derived] Chinthrajah RS, Purington N, Andorf S, Rosa JS, Mukai K, Hamilton R, Smith BM, Gupta R, Galli SJ, Desai M, Nadeau KC. Development of a tool predicting severity of allergic reaction during peanut challenge. Ann Allergy Asthma Immunol. 2018 Jul;121(1):69-76.e2. doi: 10.1016/j.anai.2018.04.020. Epub 2018 Apr 27. PMID 29709643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All arms undergo an Initial Dose Escalation (IDE) Day and updosing regimen with a maintenance phase of OIT or placebo to a maximum of 4,000 mg protein daily, as peanut flour, in the OIT groups, and to a maximum of an equivalent amount of oat flour for the placebo group.
Pre-assignment Details: At Week 104, individuals that reach criteria will, based on the randomization, either stop therapy with peanut and be switched to oat flour or will maintain on 300 mg peanut protein per day and all placebo subjects decreased to the equivalent volume of oat flour to optimize the blind. All subjects were evaluated every 13 weeks with DBPCFCs.
Groups:
- Peanut-4000: Oral immunotherapy with peanut discontinuation arm
- Peanut-300: Oral immunotherapy with low dose peanut continuation arm
- Placebo Comparator: Oat Flour 600 mg: Placebo received oat flour
Period: Overall Study
Arm/Group | Peanut-4000 | Peanut-300 | Placebo Comparator: Oat Flour 600 mg
Started | 60 | 35 | 25
Completed | 51 | 29 | 1
Not Completed | 9 | 6 | 24

BASELINE CHARACTERISTICS:
Groups:
- Peanut 4000: Oral immunotherapy with peanut discontinuation arm
- Peanut 300: Oral immunotherapy with low dose peanut continuation arm.
- Total: Total of all reporting groups
Arm/Group | Peanut 4000 | Peanut 300 | Placebo Comparator: Oat Flour 600 mg | Total
Number analyzed (Participants) | 60 | 35 | 25 | 120
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 10 [7 to 49] | 11 [7 to 47] | 11 [7 to 53] | 11 [7 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 6 | 39
  Male | 39 | 23 | 19 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 1 | 11
  Not Hispanic or Latino | 51 | 34 | 24 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 35 | 25 | 120

OUTCOME MEASURES:

1. Primary Outcome: Passing the Week 117 DBPCFC to Peanut
Description: Number of Participants with No Clinical Reactivity to Peanuts
Time Frame: Week 117 - Number of participants with no clinical reactivity to peanuts
Measure: Number; unit: participants
Arm/Group | Peanut 4000 | Peanut 300 | Placebo Comparator: Oat Flour 600 mg
Number analyzed (Participants) | 60 | 35 | 25
participants | 21 | 19 | 1

2. Secondary Outcome: Passing the DBPCFC to Peanut at Week 130
Description: Secondary endpoint: Passing the DBPCFC to peanut at 130 weeks
Time Frame: Week 130
Measure: Number; unit: participants
Groups:
- Peanut 4000: Arm A on peanut OIT until week 104 (maintenance) and once meeting criteria on OIT treatment for minimum 104 weeks, 2) taking daily maintenance dose of 4,000 mg protein for at least 13 weeks, 3) no severe reactions to home dosing from Week 91-Week 104, and 4) no reactions at the Week 104 DBPCFC] will be assigned to avoid peanut (i.e. will consume 600 mg oat flour daily) and will proceed to tolerance and desensitization phase.
  Peanut Protein 4,000mg: Arm A will be defined as "clinically tolerant" if there is no clinical reactivity at the Week 104 and Week 117 DBPCFC. Clinical reactivity is defined as any reaction ≥ Grade 1 based on the Bock's Criteria (Appendix 4). Individuals in Arm A who meet the definition of "clinically tolerant" will continue to avoid peanut protein (i.e. continue on 600 mg per day of oat flour) as long as each subsequent DBPCFC (performed every 13 weeks until end of study) shows no clinical reactivity.
  Oat Flour: Arm C will be defined as "natural l
- Peanut 300: Arm B on peanut OIT until week 104 and once meeting criteria specified in description of Arm A, will be assigned to be maintained on 300 mg peanut protein (i.e. 600 mg peanut flour) daily and will proceed to the tolerance and desensitization testing phase.
  Oat Flour: Arm C will be defined as "natural loss of responsiveness" if they show no clinical reactivity at DBPCFCs (week 117 to end of study).
  Peanut Protein 300 mg: Arm B will be defined as "desensitized" to a minimum of 300 mg per day of peanut protein if they show no clinical reactivity at DBPCFCs (week 117 to end of study).
- Placebo Comparator: Oat Flour 600 mg: Arm C that is maintained on placebo (oat flour) throughout the study; this arm will receive 600 mg oat flour beginning on week 104. This will be true even if a subject in the placebo group meets criteria at week 104
  Oat Flour: Arm C will be defined as "natural loss of responsiveness" if they show no clinical reactivity at DBPCFCs (week 117 to end of study).
Arm/Group | Peanut 4000 | Peanut 300 | Placebo Comparator: Oat Flour 600 mg
Number analyzed (Participants) | 60 | 35 | 25
participants | 12 | 15 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Description: Safety outcomes determined by Common Terminology Criteria.
Arm/Group | Peanut-4000 | Peanut-300 | Placebo Comparator: Oat Flour 600 mg
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/35 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/35 | 0/25
Other Adverse Events (participants affected / at risk) | 0/60 | 0/35 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut-4000 (N=60) | Peanut-300 (N=35) | Placebo Comparator: Oat Flour 600 mg (N=25)
eosinophilic esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — One peanut-0 participant developed eosinophilic esophagitis and his symptoms resolved after termination from the study.
anaphylaxis with moderate hypotension (General disorders) | 0 (0) | 1 (1) | 0 (0) — The other SAE occurred following an up-dosing in the peanut-300 arm. The participant engaged in vigorous exercise and experienced anaphylaxis with moderate hypotension which was reversed after one dose of injectable epinephrine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02103270/Prot_000.pdf
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT02103270/ICF_001.pdf
  • Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT02103270/SAP_002.pdf